CLINICAL TRIAL: NCT03389048
Title: Performance Assessment of the PMD-200 (Physiological Monitor Device), a Novel Pain Monitor, in Subjects With Degenerative Lumbar Spine Disease Who Requires Surgical Procedure
Brief Title: Performance Assessment Of The PMD-200 In Subjects With Degenerative Lumbar Spine Disease Who Requires Surgical Procedure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol compliance and inability to support proper performance
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLI-16-04
Record Dates: First submitted 2017-12-21; First posted 2018-01-03 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-03

CONDITIONS: Degenerative Diseases, Nervous System
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- degenerative lumbar spine disease (Experimental): patients who suffer from unilateral degenerative lumbar spine disease, undergo SLR test while being recorded by PMD-200
  Interventions: Device: PMD-200; Diagnostic Test: SLR

INTERVENTIONS:
Device: PMD-200 — The PMD-200 system is comprised of a console and designated finger probe with 4 sensors. The Sensors are Photoplethysmography (PPG) Galvanic Skin Response (GSR), Accelerometer (ACC) and Thermistor (TMP)
Diagnostic Test: SLR — With the patient lying down on his/her back, the examiner lifts the patient's leg while the knee is straight.

SUMMARY:
Performance assessment of the PMD-200, a novel pain monitor, in subjects with degenerative lumbar spine disease who requires surgical procedure

DETAILED DESCRIPTION:
The proposed study is design to further demonstrates the capability of the Nociception Level, (NoL) Index in identify and discriminate between painful event and non-painful period following pain stimulus of Straight Leg Raising (SLR) test in patients with degenerative lumbar spine disease. This feasibility study may provide first indication for a validation method that will be able to evaluate the outcome of a surgical procedure within the degenerative lumbar spine patient. Currently, there is lack of understanding of long-term outcomes after such surgeries.

In this study, the investigators plan to demonstrate that the NoL Index may serve as an indicator to the surgical procedure outcome. It will compare the objective measurement of the NoL to the patient Visual Analogue Scale (VAS) score and disability questionnaire that will characterize the subject pain perception prior and following the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 and less than 65 (18 < Age < 65).
* The subject suffer from unilateral degenerative lumbar spine disease
* The subject suffer from leg pain only in one leg, while no pain in the other leg.
* The subject was hospitalized in the neurosurgery department of the hospital in order to undergoes spinal surgery due to the above disease
* A signed Informed Consent Form (ICF) has been obtain from the subject

Exclusion Criteria:

* The subject has a bi-lateral degenerative lumbar spine disease
* The subject is pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
discrimination between nonpainful period to painful period | Through study completion, about one year
  To demonstrate that the NoL index can discriminate between nonpainful period to painful period, prior and following SLR test

SECONDARY OUTCOMES:
Correlates with changes in pain levels | Through study completion, about one year
  To demonstrate that the NoL Index is correlates with changes in pain levels of the subject prior and following SLR.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Soustiel, Prof., Principal Investigator — Dept. of Neurosurgery Galilee Medical Center, Nahariya, Israel
Locations (1):
- Galil Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No